CLINICAL TRIAL: NCT00987896
Title: A Novel Endoscopic Device (Megachannel™) For Repeated Right Colonic Access During Colonoscopy
Brief Title: Megachannel Device for Advanced Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Arnulf Ferlitsch, MD, Medizinische Universität Wien
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: megachannel
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Multiple Polyps Right Colon; Large Polyp Right Colon; Suspected Polyp Right Colon
Keywords: colonoscopy; polypectomy; NOTES
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Megachannel Application (Experimental): Colonoscopy with loaded Megachannel is performed
  Interventions: Device: Colonoscopy with Megachannel™ device loaded

INTERVENTIONS:
Device: Colonoscopy with Megachannel™ device loaded — Before colonoscopy, megachannel is loaded on the endoscope, during colonoscopy megachannel will be inserted into the patient via the endoscope placed in the colon
  Other Names: Megachannel(TM), produced by Minos Medical, Irvine, CA

SUMMARY:
Megachannel is a newly developed colonic access system allowing rapid and multiple passes of the colonoscope to the right colon.

The investigators want to conduct a multinational study to evaluate the safety and clinical feasibility of placing a 100 cm Megachannel prototype in the right colon.

DETAILED DESCRIPTION:
Patients scheduled for colonoscopy with suspected right colonic polypoid lesions will be included. The prototype will loaded onto a 160 cm lower GI endoscope and introduced via colonoscopic guidance. Time to cecum, total investigation time, clinical feasibility and complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for colonoscopy with suspected large or multiple polys in the right colon

Exclusion Criteria:

* previous abdominal surgery
* history or currently diagnosed intra-abdominal cancer
* patients presenting with unstable angina
* drug abusers
* pregnant women
* patients with known colonic strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety and clinical feasibility of performing colonoscopy with megachannel | during every single colonoscopy in the study

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Silberhumer GR, Birsan T, Noda W, Unger E, Mayr W, Lang S, Prager G, Gasche C. Design and instrumentation of new devices for performing appendectomy at colonoscopy (with video). Gastrointest Endosc. 2008 Jul;68(1):139-45. doi: 10.1016/j.gie.2008.02.024. Epub 2008 May 2. PMID 18455170
- [Derived] Ferlitsch A, Silberhumer GR, Noda W, Birsan T, Desai D, Kumar A, Rao GV, Khakar A, Gomez NA, Gasche C. A novel endoscopic device for repeated right-side colonic access during colonoscopy (with video). Gastrointest Endosc. 2010 May;71(6):1052-5. doi: 10.1016/j.gie.2009.12.059. PMID 20438892